CLINICAL TRIAL: NCT06711432
Title: Effects of Different Intraoperative Blood Pressure Management Strategies on Postoperative Cognitive Function and Adverse Outcomes in Tumor Patients With High Risk Factors for Stroke
Brief Title: Different Intraoperative Blood Pressure Management on Postoperative Cognitive Function in Tumor Patients（PRECISION）
Acronym: PRECISION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhu Yejing, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-2024-556
Record Dates: First submitted 2024-08-10; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Tumor; Stroke
Keywords: blood pressure management strategies; postoperative cognitive function; tumor patients; high risk factors for stroke
MeSH Terms: conditions — Neoplasms; Stroke | interventions — Norepinephrine; Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strict Blood Pressure Management Group (MAP > 80 mmHg) (Experimental): Management strategy: For patients assigned to strict blood pressure management, stop taking ACEI (angiotensin converting enzyme inhibitors) or ARB (angiotensin receptor blockers) on the day of surgery. Other antihypertensive drugs can be given selectively depending on the patient's blood pressure level. Intraoperative use of norepinephrine or phenylephrine (norepinephrine 0.01-0.1μg/kg/min or phenylephrine 0.15-1.1 ug/kg/min). The actual infusion speed depends on achieving the target MAP.
  Interventions: Drug: Norepinephrine or phenylephrine
- Management strategy of the conventional blood pressure management group (MAP>65mmHg (No Intervention): For patients assigned to the conventional blood pressure management group, ACEI, ARB or calcium antagonists can be used until the morning of the day of surgery if the anesthesiologist deems it necessary. Intraoperative blood pressure management is based on routine, and it is not necessary to use pressor drugs prophylactically, which can be used according to the actual clinical situation. In general, intraoperative MAP should not be lower than 65mmHg. If there is no contraindication of hypotension, oral antihypertensive drugs can be resumed as soon as possible after surgery.

INTERVENTIONS:
Drug: Norepinephrine or phenylephrine — Intraoperative use of norepinephrine or phenylephrine (norepinephrine 0.01-0.1ug/kg/min, or phenylephrine 0.15-1.1 ug/kg/min). The actual infusion speed depends on reaching the target MAP(>=80mmHg).
  Arms: Strict Blood Pressure Management Group (MAP > 80 mmHg)

SUMMARY:
This is a randomized controlled study to explore whether perioperative blood pressure management with different strategies can reduce the incidence of delirium and postoperative cognitive impairment and serious perfusion related complications (persistent hypotension, new heart arrhythmia, cardiac insufficiency, new stroke, sudden death, etc.) within 30 days after stroke in cancer patients at high risk for stroke.

Patients were randomly divided into: 1) strict blood pressure management group: norepinephrine or phenylephrine maintenance intraoperative MAP≥85 mmHg, and 2) conventional blood pressure management group: intraoperative routine blood pressure management (MAP≥65mmHg).

The study included 424 subjects and was randomized to provide 90% efficacy. Secondary markers were unscrupulous cerebrovascular events (persistent hypotension, arrhythmia, cardiac insufficiency, new stroke, sudden death) within 30 days after surgery.

DETAILED DESCRIPTION:
After entering the operating room, invasive blood pressure, heart rate, electrocardiogram and SpO2 were monitored, central vein was opened, and intravenous administration of Sufentanil 0.3-0.5ug/kg, etomidate 0.3mg /kg and rocurobromide 0.9mg/kg were performed after induction of anesthesia. Mechanical ventilation, VT 6-8 mL/ kg, RR 12-16 times/min, PETCO2 3540mmHg maintained. Intraoperative continuous infusion of propofol and remifentanil to maintain Bis 40-60 (TCI or constant velocity?) . Do not use dexmedetomidine or benzodiazepines during anesthesia; Scopolamine and penehyclidine are also prohibited because they promote the occurrence of postoperative delirium. Atropine is only used to treat bradycardia when necessary. The MAP set threshold is maintained in the two groups of patients, below the threshold, as follows: 1. Administer reasonable vasoactive drugs, and record the dose; 2. Appropriate fluid infusion and body position changes are given and recorded; 3. Intraoperative blood gas analysis was monitored to maintain electrolyte homeostasis; 4. Once the hematocrit is less than 28%, give blood transfusion; 30 minutes before the end of surgery, 0.1-0.2ug/kg sufentanil was used as analgesic load. Peripheral nerve blocks, such as paravertebral block, transverse abdominal muscle plane block, etc., or combined epidural anesthesia are routinely performed.

Patients without contraindications were routinely given an NSAID-type drug combined with acetaminophen (acetaminophen 500mg or flurbiprofen 50mg or parexib 40mg) before incision. According to clinical routine infusion, blood transfusion/blood products if necessary, maintain urine volume >0.5ml/kg/h, hemoglobin ≥8g/dL. During the operation, the nasopharyngeal temperature was maintained at 36-37C.

Treatment after operation: The patient was admitted to the postoperative recovery room (PACU) after the operation and recovery and extubation, or entered the PACU with tube; Routine monitoring includes non-invasive blood pressure, pulse oxygen saturation and electrocardiogram. Stay at PACU for at least 30 minutes and return to the ward after the modified Aldrete score is ≥9. Unstable patients are sent to the ICU after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high-risk stroke (combined with 3 risk factors or more according to the stroke risk screening table)
2. Patients who plan to undergo surgery for abdominal tumors (gynecological, urinary, hepatobiliary, and gastrointestinal tumors) under general anesthesia are expected to have surgery duration >2 hours
3. The ASA is rated as Class II or III
4. Patients who underwent invasive arterial blood pressure monitoring before surgery signed informed consent

Exclusion Criteria:

1. Patients do not want to participate in the study
2. Patients with severe heart disease (severe valvular disease, sick sinus syndrome, high atrioventricular block without pacemaker implantation), grade III or above Liver function impairment (Child-Pugh class C)
3. Need kidney replacement therapy; New stroke <3 months
4. Emergency surgery
5. Preoperative history of mental illness, epilepsy, Parkinson's disease, or myasthenia gravis
6. Speech, vision, or hearing impairment that prevents completion of a cognitive function assessment
7. Situations where strict blood pressure management is not appropriate, such as controlled hypotension during surgery.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative delirium and cognitive function in patients with high-risk stroke. | in one week after surgery
  We use the Consciousness Ambiguity Measure (CAM) for POD assessment at 3, 5, and 7 days postoperatively. The 3-Minute Confusion Assessment Measure (3D-CAM) is used for POD assessment at 3, 5, and 7 days postoperatively, and the Memory Confusion Assessment Scale (MDAS) is used for POD severity scoring. Scores are taken twice, at 10:00 am and 5:00 pm, and are assessed by trained researchers (non-anesthesia personnel) who conduct cognitive tests. If a patient experiences an acute change or fluctuation in their mental state, decreased attention, confusion of thought, or a change in level of consciousness, then delirium is present. If delirium requires intervention, the patient receives an intravenous injection of haloperidol, and if necessary, it is repeated every 60 minutes and recorded promptly.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 30 days after surgery.
  Adverse cardiovascular events within 30 days after surgery were recorded: Such as persistent hypotension, arrhythmia, heart failure, and new strokes. Record the incidence of complications (new conditions that require medical intervention) within 30 days after surgery (including the hospitalization period) (follow-up by phone for discharged patients) postoperative survival status.

OTHER OUTCOMES:
S100 calcium-binding protein B | on postoperative day 3 and one week after surgery
  S100B was measured using the enzyme-linked immunosorbent assay (ELISA) (Merck & Co Inc, USA) according to manufacturer's instructions.
BDNF | on postoperative day 3 and one week after surgery
  BDNF was measured using the enzyme-linked immunosorbent assay (ELISA) (Merck & Co Inc, USA) according to manufacturer's instructions.
ubiquitin C-terminal hydrolase-L1 (UCH-L1) | on postoperative day 3 and one week after surgery
  UCH-L1 was measured using the enzyme-linked immunosorbent assay (ELISA) (Merck & Co Inc, USA) according to manufacturer's instructions.
neurofilament light chain protein (NfL) | on postoperative day 3 and one week after surgery
  NfL was measured using the enzyme-linked immunosorbent assay (ELISA) (Merck & Co Inc, USA) according to manufacturer's instructions.
cardiac troponin I | on postoperative day 3 and one week after surgery
  cardiac troponin I was measured using the enzyme-linked immunosorbent assay (ELISA) (Merck & Co Inc, USA) according to manufacturer's instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China